CLINICAL TRIAL: NCT04645641
Title: Evaluation of the Safety and Effectiveness of the Dexcom Glucose Monitoring (CGM)
Brief Title: Evaluation of the Safety and Effectiveness of the Dexcom Glucose Monitoring (CGM) System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PTL-904120
Record Dates: First submitted 2020-11-02; First posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Masking Description: All systems worn will be blinded. Sensor wear locations will be pre-assigned. All sensor insertions will be performed at the clinic by study staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CGM Users (Active Comparator): Glucose challenge during clinic sessions to assess performance of CGM compared to comparator measurement.
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Continuous Glucose Monitoring System

SUMMARY:
Evaluation of the Safety and Effectiveness of the Dexcom Glucose Monitoring (CGM) System

DETAILED DESCRIPTION:
The objective of the study is to establish performance of the Dexcom CGM System (System) in comparison to a blood glucose comparator method.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 or older
* Diagnosis of Type 1 diabetes or Type 2 diabetes
* Willing to wear the required number of Systems for the total duration of study wear
* Willing to participate in Clinic Session(s) during study wear

Exclusion Criteria:

* Presence of extensive skin changes/diseases at sensor wear site(s) that preclude wearing the sensor(s) on skin
* Known allergy to medical-grade adhesives
* Pregnancy
* Hematocrit outside specification
* ≥ 18 years of age:

  * Male: 36.0%;
  * Female: 33.0%;
* 13-17 years of age: 35.0%;
* 7 years - 12 years of age: 32.0%;
* End stage renal disease and currently managed by dialysis or anticipating initiating dialysis during the study wear period
* Required or scheduled to have a Magnetic Resonance Imaging (MRI) scan, Computed Tomography (CT) scan, or diathermy during the study wear period

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-10-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
System Performance | 10 days
  System Performance will be characterized with respect to comparator venous plasma measurements.

SECONDARY OUTCOMES:
System Related Adverse Device Effects | 10 days
  System will be characterized by Adverse Device Effects experienced by study participants

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - AMCR Institute, Escondido, California
  - Barbara Davis Center, Aurora, Colorado
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Endeavor Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No